CLINICAL TRIAL: NCT00176956
Title: Atopic Dermatitis-Like Skin Disease in Pediatric Heart Transplant Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IRB approval has lapsed.
Sponsor: Hordinsky, Maria K., MD (Individual)
Responsible Party: Sponsor
Organization: University of Minnesota (Other)
Other Study IDs: 0110M09983
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Dermatitis
Keywords: Post Pediatric Heart Transplant
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Skin Biopsy — Skin biopsy.
  Other Names: Skin biopsy.

SUMMARY:
The skin disease found in pediatric heart transplant patients represents an atopic dermatitis-like rash that is refractory to systemic immunomodulation.

DETAILED DESCRIPTION:
We want to determine whether pediatric heart transplant patients with an atopic dermatitis-like rash report a personal and/or family history of atopy (asthma, allergies and atopic dermatitis). In addition comparisons will be made between the presence of atopy between patients with and without the skin rash. Comparisons will be made of systemic immunosuppressive therapies between patients with and without the atopic dermatitis-like rash. Determination will be made as to whether histologic characterization of a skin biopsy specimen is consistent with AD. Thorough evaluations will be made of patients in the clinic with this rash and the presence of bacterial superinfection will be ruled out.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had a heart transplant.
* Patients must be less than 16 years of age.

Exclusion Criteria:

* Patients who have not had a heart transplant.
* Patients who are greater than 16 years of age.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2002-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States